CLINICAL TRIAL: NCT02206659
Title: An Open-label Evaluation of Trough and Peak Effects of 40 mg Telmisartan Tablet by Ambulatory Blood Pressure Monitoring in Chinese Patients With Mild to Moderate Essential Hypertension
Brief Title: Effects of Telmisartan by Ambulatory Blood Pressure Monitoring (ABPM) in Chinese Patients With Mild to Moderate Essential Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 502.367
Record Dates: First submitted 2014-07-31; First posted 2014-08-01 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2014-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan

ARMS (1):
- Telmisartan (Experimental): 2-week placebo run-in period followed by 6 weeks of treatment with telmisartan
  Interventions: Drug: Telmisartan; Drug: Placebo

INTERVENTIONS:
Drug: Telmisartan
Drug: Placebo

SUMMARY:
To assess the trough/peak ratio of 40 mg Telmisartan tablet by ambulatory blood pressure monitoring in Chinese patients with mild to moderate essential hypertension

ELIGIBILITY:
Inclusion Criteria:

* Chinese male or female aged 18 to 75 years
* Mild to moderate hypertension defined as a morning DBP _95 and <110 mm Hg at visit1 and visit 2. Mean sitting systolic pressure (SBP) must be <180 mm Hg
* Ability to provide written informed consent

Exclusion Criteria:

* Women who are pregnant or breast-feeding, or of childbearing potential without an effective method of birth control (effective birth control methods are: uterine device, surgical sterilisation, progestogens alone)
* Known or suspected secondary hypertension
* Known history of any chronic hepatic disease
* Bilateral renal artery stenosis; renal artery stenosis in a solitary kidney; post-renal transplant
* New York Heart Association (NYHA) functional class congestive heart failure (CHF) III-IV
* Unstable angina pectoris
* Myocardial infarction or percutaneous transluminal coronary angiography (PTCA) or cardiac surgery within the preceding three months
* Clinical relevant cardiac arrhythmias as determined by the clinical investigator
* Hypertrophic obstructive cardiomyopathy or clinically significant valvular disease
* Evidence of retinal hemorrhages/exudates
* Clinical significant hyperkalemia as defined by serum potassium level >6.0 milliequivalents (mEq)/L
* Insulin-dependent diabetes mellitus
* Non-insulin-dependent diabetes mellitus with poor glucose control as defined by persistent fasting blood sugar >200 mg/dl, peripheral neuropathy or autonomic neuropathy
* Known drug or alcohol dependency
* Administration of any diuretic, ACE inhibitor or angiotensin II receptor antagonist within two weeks before run-in period
* Administration of medication known to affect blood pressure during trial period
* Patients receiving any investigational therapy within one month of signing the informed consent form
* Known hypersensitivity to any component of the formulation
* Any other clinical condition which, in the opinion of the principal investigator, would not allow safe completion of the protocol and safe administration of trial medication

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2000-08; Primary Completion 2001-02 (Actual)

PRIMARY OUTCOMES:
Mean of trough/peak (T/P) ratio for diastolic blood pressure (DBP) and systolic blood pressure (SBP) | 42 days after start of treatment
Median of T/P ratio for DBP and SBP | 42 days after start of treatment

SECONDARY OUTCOMES:
Change in mean 24-hr DBP and SBP | Day -13, 42 days after start of treatment
Change in daytime mean for SBP and DBP | Day -13, 42 days after start of treatment
Change in nighttime mean for SBP and DBP | Day -13, 42 days after start of treatment
Change in mean of DBP and SBP for last 6-hr dosing interval | Day -13, 42 days after start of treatment